CLINICAL TRIAL: NCT03322878
Title: Intravenous Versus Caudal Magnesium Sulfate as an Adjuvant to Caudal Bupivacaine in Lower Abdominal Surgeries in Paediatrics Under General Anaesthesia
Brief Title: Magnesium Sulfate as an Adjuvant to Caudal Bupivacaine in Lower Abdominal Surgeries in Paediatrics.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Magda saleh rezk, Assistant lecturer, anesthesia department,Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: N-45 -2017
Record Dates: First submitted 2017-10-24; First posted 2017-10-26 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Pain, Postoperative
Keywords: postoperative pain , pediatrics , magnesium sulfate
MeSH Terms: conditions — Pain, Postoperative | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intravenous magnesium group (Group IV) (Experimental): Group IV (n=30) will receive intravenous (IV) 20 ml magnesium SO4 (50 mg/ kg 10% MgSO4(magnesium sulphate) diluted in normal saline to a total volume of 20 ml(milliliter) ) and caudal anaesthesia using (bupivacaine 0.25% diluted in normal saline with total volume of 1 mL/kg) .
  Interventions: Drug: Magnesium SO4
- Caudal magnesium group (Group CA) (Active Comparator): Group CA (n=30) will receive IV 20 ml normal saline and caudal anaesthesia using (bupivacaine 0.25% and 50 mg Magnesium SO4 diluted in normal saline with total volume of 1mL/kg).
  Interventions: Drug: Magnesium SO4
- Placebo group (Group P) (Placebo Comparator): Group P (n=30) ) will receive IV 20 ml normal saline and caudal anaesthesia using (bupivacaine 0.25% diluted in normal saline with total volume of 1 mL/kg).
  Interventions: Drug: Magnesium SO4

INTERVENTIONS:
Drug: Magnesium SO4 — The intravenous solutions (magnesium 10% for group IV or saline 0.9% for group CA and P) will be started then caudal block will be performed by the same anesthetist. Under complete aseptic conditions a caudal puncture with 5 cm short beveled 22 G caudal needle will be used in the lateral decubitus position. After identifying the space using the loss of resistance technique with saline, the study solutions will be injected slowly with repetitive intermittent aspiration.
  Other Names: Caudal anaesthesia

SUMMARY:
Intravenous magnesium has been studied in pediatrics to reduce agitation after sevoflurane anesthesia in children undergoing adenotonsillectomy, reduce intraoperative rocuronium requirements, prevent laryngospasm and coughing after removal of the endotracheal tube in patients undergoing adenotonsillectomy.

The aim of this study is to investigate the role of intravenous magnesium sulfate on postoperative pain management in paediatrics and to compare it with its effect when administered caudally in children undergoing lower abdominal surgeries.

DETAILED DESCRIPTION:
Postoperative pain in children is difficult to assess and is associated with strong emotional component .

Recently, there is an increasing interest to study magnesium analgesic effects. Magnesium, the fourth most common cation in the body, inhibits calcium entry into the cell via a noncompetitive blockade of the N-methyl-d-aspartate (NMDA) receptors. Magnesium and the NMDA receptors are thought to be involved in the modulation of pain. Magnesium is also a physiological calcium antagonist at different voltage-gated channels, which may be important in the mechanisms of antinociception.

As a NMDA antagonist, magnesium prevents the central sensitization from nociceptive stimulation. Many studies suggested that epidurally administered magnesium as an adjuvant could reduce the postoperative pain in adults. But few studies are available about the use of magnesium as an adjuvant in caudal block for postoperative analgesia in pediatrics.

The aim of this study is to investigate the role of intravenous magnesium sulfate on postoperative pain management in paediatrics and to compare it with its effect when administered caudally in children undergoing lower abdominal surgeries.

Objectives

1. To determine the analgesic effect of intravenous magnesium in children undergoing lower abdominal surgeries.
2. To evaluate and compare the efficacy of magnesium sulfate when administered intravenously versus caudally.
3. To evaluate the sedative effect of intravenous magnesium in paediatrics.
4. To illustrate the role of hypomagnesemia in post-operative pain.

Population of study & disease condition Paediatric patients undergoing lower abdominal surgeries.

Methodology in details Patients fulfilling the study inclusion criteria will be recruited and enrolled in the study after Ethical Committee approval. All parents will sign an informed consent to participate in the study after detailed explanation of the expected benefits and possible risks.

Study groups This study will be performed in Cairo University specialized pediatric Hospital after approval of the Research Ethical Committee, and written informed consents from the parents.

90 participants will be randomly assigned using an online randomization program (http://www.randomizer.org) and the sealed envelop method into three groups:

1. Intravenous magnesium group (Group IV)
2. Caudal magnesium group (Group CA)
3. Placebo group (Group P).

Preoperative assessment:

History taking, clinical examination and routine laboratory investigations will be checked for all patients to exclude any of the above mentioned exclusion criteria.

Intraoperative management:

After arrival of the patient to the operating theater 5 leads electrocardiography (ECG), automated non-invasive blood pressure monitoring (NIBP) and a pulse oximetry will be applied. Anaesthesia will be induced by inhalation of 6- 8 % sevoflurane , by an anesthetist blinded to the group allocation. Once consciousness is lost , intravenous access will be established, fentanyl (1- 2 μg/kg ) and atracurium (0.5 mg/ kg) will be given to facilitate tracheal intubation. Anaesthesia will be maintained by 1.2 % isoflurane, atracurium top up doses under controlled ventilation.

The intravenous solutions (magnesium 10% for group IV or saline 0.9% for group CA and P) will be started then caudal block will be performed by the same anesthetist. For caudal puncture a 5 cm short beveled 22 G caudal needle will be used in the lateral decubitus position. After identifying the space using the loss of resistance technique with saline, the study solutions will be injected slowly with repetitive intermittent aspiration. Rescue analgesia in the form of fentanyl 1 μg/kg will be administered if haemodynamic parameters (blood pressure and heart rate) increased 20 % from the baseline.

Surgery will be allowed to begin 10 min after performing the block. After emergence from anaesthesia, patients will be managed by an observer blinded to group allocation in the post anaesthesia care unit (PACU). Postoperative rescue analgesia in the form of rectal paracetamol (80-120mg) if pain score (Children's Hospital of Eastern Ontario Pain Scale CHEOPS was > 8 to be repeated every 6 hours if needed not to exceed 5 doses / 24 hr.

Statistical analysis:

SPSS(Statistical Package for Social Sciences) version 20.0 will be used for data entry and data management. Mean ± standard deviation will describe quantitative variables and proportions for qualitative variables. ANOVA with mixed model will be used to show time effect (e.g change of pain score over time post-operatively) and to show group effect, (compare rate of change among 3 study groups). P value will be set significant at 0.05 level and always 2 tailed.

Sample size (number of participants included) This study hypothesized that at least 2 of the 3 study groups are significantly different regarding pain score after 6 hours post-operatively.With a type I error of 0.05, power of a test of 0.90 and a difference to be detected in pain score of 1.3 with background standard deviation of 0.9 (based on results from a study by H.-S. Na, J.-H. Lee, J.-Y. Hwang, J.-H. Ryu, S.-H. Han, Y.-T. Jeon and S.-H. Do.Effects of magnesium sulphate on intraoperative neuromuscular blocking agent requirements and postoperative analgesia in children with cerebral palsy.British Journal of Anaesthesia 104 (3): 34450(2010)doi:10.1093/bja/aep379& Gamal T. Yousef, Tamer H. Ibrahim, Ahmed Khder, et al. Enhancement of ropivacaine caudal analgesia using dexamethasone or magnesium in children undergoing inguinal hernia repair. Anesth Essays Res. 2014 Jan-Apr; 8(1): 13-19. doi: 10.4103/0259-1162.128895 , which showed a mean score of 2.4±0.9 in caudal group with IV magnesium versus 3.7±0.9 in control group), at least 16 patients per group is needed. To warrant normal distribution of study variables a total of 90 patients will be recruited in this study who will be randomized into 30 patient per group .

ELIGIBILITY:
Inclusion Criteria:

* age between 1 and 7 years, ASA(American Society of Anesthesiologists) physical status class |- || , patients scheduled for lower abdominal surgeries.

Exclusion Criteria:

* patients with psychiatric disorders , children with cardiovascular,respiratory ,hepatic or renal dysfunction , known contraindications to regional anesthesia, ASA class |||- |V, hypersensitivity to magnesium or regular analgesic drugs.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The analgesic effect of intravenous magnesium in children undergoing lower abdominal surgeries | 12 hours
  Post operative pain score will be assessed using children's Hospital of Eastern Ontario Pain scale which is based on 6 criteria:
  * Crying
  * Facial expression
  * Child verbal expression
  * Torso (body position)
  * Touching or grabbing at wound
  * Legs position Criterion 1 is given a score of 1-3, criterion 2 and 3 are given a score of 0-2 while criterion 4, 5 and 6 are given a score of 1-2; making the worst possible score 13 while the least possible score is 4. A total score ≤ than 8 indicate adequate analgesia.

SECONDARY OUTCOMES:
Time to first rescue analgesia | 12 hours
  Post operative first rescue analgesia time
Post operative sedation score | 30 minutes
  Sedation will be monitored after PACU arrival using Ramsay score : 1=fully awake , 2=drowsy but awakens spontaneously , 3=asleep but arouses and responds appropriately to simple verbal commands , 4=asleep,unresponsive to commands,but arouses to shoulder tap or loud verbal stimulus , 5=asleep and only responds to firm

CONTACTS AND LOCATIONS:
Overall Officials: Manal M El gohary, Principal Investigator — Professor; Amina A Ela, Study Director — Assistant professor; Heba M Nassar, Study Chair — Assistant professor